CLINICAL TRIAL: NCT02800811
Title: Randomized, Double-blind, Placebo-controlled, Dose-escalation Study for the Assessment of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Intravenous Doses of FR104 in Healthy Subjects
Brief Title: Safety, Tolerability, PK, PD, and Immunogenicity of Single and Multiple Ascending Intravenous Doses of FR104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FR104-CT01; 2015-000302-19 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-06-15 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis; Complication of Transplant
Keywords: FR104; CD28; immunomodulation; T regulatory cell; Pegylated monovalent anti-CD28 Fab antibody
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Part 1: Cohort A, Group 1, FR104 (Experimental): Dose: single 0.005 mg/kg.
  Interventions: Drug: FR104
- Part 1: Cohort A, Group 2, FR104 (Experimental): Dose: single 0.05 mg/kg.
  Interventions: Drug: FR104
- Part 1: Cohort A, Group 3, FR104 (Experimental): Dose: single 0.2 mg/kg.
  Interventions: Drug: FR104
- Part 1: Cohort A, Group 4, FR104 (Experimental): Dose: single 0.5 mg/kg.
  Interventions: Drug: FR104
- Part 1: Cohort A, placebo (Placebo Comparator): Placebo, single administration, double blind (1/4 healthy subject in group 1, 1/4 in group 2, 2/5 in group 3 and 2/5 in group 4).
  Interventions: Drug: Placebo
- Part 1: Cohort B, Group 7, FR104 (Experimental): Dose: single 0.5 mg/kg. Healthy subject naïve to KLH and that will receive a KLH challenge.
  Interventions: Drug: FR104
- Part 1: Cohort B, Group 8, FR104 (Experimental): Dose: single 0.2 mg/kg. Healthy subject naïve to KLH and that will receive a KLH challenge.
  Interventions: Drug: FR104
- Part 1: Cohort B, Group 9, FR104 (Experimental): Dose: single 1.5 mg/kg. Healthy subject naïve to KLH and that will receive a KLH challenge.
  Interventions: Drug: FR104
- Part 1: Cohort B, Group 9 bis, FR104 (Experimental): Dose: single 0.02 mg/kg group. Healthy subject naïve to KLH and that will receive a KLH challenge.
  Interventions: Drug: FR104
- Part 1: Cohort B, placebo (Placebo Comparator): placebo, single administration, double-blind: healthy subjects naïve to KLH and that will receive a KLH challenge (2/5 in each group of cohort B)
  Interventions: Drug: Placebo
- Part 2: Group 10, FR104 (Experimental): Dose: repeat, 0.2 mg/kg. Two administrations separated by an interval of 28 days.
  Interventions: Drug: FR104
- Part 2: Group 11, FR104 (Experimental): Dose: repeat, 0.5 mg/kg. Two administrations separated by an interval of 28 days.
  Interventions: Drug: FR104
- Part 2: placebo (Placebo Comparator): placebo, repeat, double-blind: 2/5 subjects in each group of Part 2. Two administrations separated by an interval of 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FR104 — GMP FR104 is provided to the site in extractable volume vials containing FR104. Appropriate Dilutions in Ringer's lactate solution is made on site.
  Arms: Part 1: Cohort A, Group 1, FR104; Part 1: Cohort A, Group 2, FR104; Part 1: Cohort A, Group 3, FR104; Part 1: Cohort A, Group 4, FR104; Part 1: Cohort B, Group 7, FR104; Part 1: Cohort B, Group 8, FR104; Part 1: Cohort B, Group 9 bis, FR104; Part 1: Cohort B, Group 9, FR104; Part 2: Group 10, FR104; Part 2: Group 11, FR104
Drug: Placebo — The placebo injection contains the vehicle. For placebo dosing, vehicle is administered in accordance with the volume of study drug administered.
  Arms: Part 1: Cohort A, placebo; Part 1: Cohort B, placebo; Part 2: placebo

SUMMARY:
First-in-human, phase I, randomized, double-blind, placebo-controlled, single center study evaluating single and multiple ascending intravenous doses of FR104 in healthy subjects.

DETAILED DESCRIPTION:
This study is a first-in-human, phase I, randomized, double-blind, placebo-controlled, single center study evaluating single and multiple ascending intravenous doses of FR104 in healthy subjects.

64 healthy male and female subjects are selected according to the inclusion and exclusion criteria, i.e., 50 subjects in Part 1 (SAD: 2 cohorts of 22 [Cohort A], 28 [Cohort B], respectively) and 14 subjects in Part 2 (MAD). The total duration of the study is 10 months.

All FR104 doses are administered intravenously by a slow infusion of at least 30 minutes. A staggered approach is observed within all dose levels. An interval of at least 14 days (last to first administration) is observed between all dose levels. Individual subjects on a same day of dosing are dosed at least 60 minutes apart.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria are eligible to participate in this study:

1. Male or female, aged 18 to 60 years, extremes includes;
2. In good health condition [medically stable] as determined on the basis of medical history, vital signs, clinical laboratory testing, and general physical examination performed at screening; Note: a retest can be done in case of an out of range clinical laboratory test value that will determine a subject's eligibility. This retest is preferably to be done at an unscheduled visit. The result of the retest are considered for subject eligibility. If the retest is outside normal reference ranges, the subject are eligible for inclusion only if the investigator judges the abnormalities to be not clinically significant.
3. Electrocardiogram (ECG) within normal range, or showing no clinically relevant deviations, as judged by the investigator; Note: a retest can be done in case of an out of range ECG value that can determine a subject's eligibility.
4. Weighs at least 50 kg and no more than 100 kg and has a Body Mass Index (BMI) within normal range: 18.0≤BMI<30.0 kg/m2;
5. Negative urine test for selected drugs of abuse at screening;
6. Negative alcohol breath test at screening;
7. Female subject is postmenopausal or surgically sterile (having had a hysterectomy, bilateral oophorectomy, or tubal ligation);
8. Female subject has a negative pregnancy test at screening;
9. Non-vasectomized male subjects having a female partner of childbearing potential must agree to the use of an effective method of contraception until 90 days after the last administration of study drug ;
10. Male subject has to agree not to donate sperm until 90 days after the last administration of study drug;
11. Willing to adhere to the prohibitions and restrictions specified in this protocol;
12. Informed Consent Form (ICF) signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study;
13. Subjects were to be EBV-positive as per positive IgG Epstein-Barr nuclear antigen (EBNA) test;
14. Nonsmoker or light smoker, i.e., smokes maximal 5 cigarettes (or 3 cigars or 3 pipe-full) per day, and ability and willingness to refrain from smoking during confinement and ambulant visits in the clinical research center.

    For Part 1, Cohort B only:
15. The subject did not undergo a KLH challenge.

Exclusion Criteria:

Subjects meeting one or more of the following criteria are excluded from participation in this study:

1. A history of any clinically significant (as determined by the investigator) cardiac, endocrinology, hematology, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy excluding non-melanoma skin cancer;
2. A known allergy, hypersensitivity, or intolerance to the study drug, or to any of its compounds;
3. The subject has a history of severe allergic or anaphylactic reactions;
4. The subject has a history of consuming more than 21 (14 for females) units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 330 mL of beer, 110 mL of wine or 28 mL of spirits);
5. Evidence or history of any clinically significant infections within the past 3 months;
6. History of or evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB) diagnosed by a positive QuantiFERON® TB-Gold In Tube test or a positive tuberculin skin test ("Mantoux") in case of a weak positive QuantiFERON® TB-Gold In Tube test;
7. Subjects with known clinically relevant immunological disorders, or auto-immune disorders, (e.g., rheumatoid arthritis, lupus erythematosus, scleroderma, etc...);
8. Subjects with a recent infection of EBV diagnosed by a positive IgM VCA;
9. A positive hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV] antibodies [Abs]) or positive human immunodeficiency virus (HIV) antibody screens;
10. The subject has a supine systolic blood pressure (SBP) <90 or >160 mmHg and a diastolic blood pressure (DBP) <50 or >90 mmHg, or pulse rate higher than 100 bpm, either at screening (blood pressure measurements taken after subject has been resting in a supine position for a minimum of 5 minutes); Note: a retest can be done in case of an out of range vital signs value that will determine a subject's eligibility. The result of the retest are considered for subject eligibility.
11. The subject is pregnant or breastfeeding;
12. The subject has received a vaccine within 60 days prior to study drug administration;
13. The subject has received any systemic immunosuppressant agent within 6 months prior to study drug administration;
14. The subject has received any antibody or biologic medicinal product within 6 months prior to study drug administration;
15. The subject has received any systemic steroid within 2 months prior to study drug administration;
16. Use of a prohibited therapy within 14 days prior to study drug administration;
17. Receipt of any investigational drug within 30 days or ten half-lives, whichever is longer, prior to the initial study drug administration;
18. The subject is participating in another clinical trial or has participated in another dose group of the current trial;
19. Had a significant blood loss (including blood donation [>500 mL]) or having had a transfusion of any blood product within the 60 days or donated plasma within 7 days prior to the initial study drug administration;
20. A condition that, in the opinion of the investigator, could compromise the well-being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements.
21. Intent to visit regions where tuberculosis and mycosis are endemic during the period of 3 months after dosing (4 months after dosing for subjects in Cohort C) , i.e., deserts areas, Eastern Europe, Central and South America, Africa except Egypt, Russia, Asia, Indonesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, timing, seriousness and relatedness of treatment emergent adverse events, and abnormalities in laboratory parameters in healthy volunteers of FR104 compared to placebo after single (SAD) and two IV doses (MAD). | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.

SECONDARY OUTCOMES:
Area under the concentration time curve to last quantifiable concentration [AUC (0-T)] after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Terminal half-life (T1/2) of FR104 after single and two repeat iv administrations | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Durations of 100%, 50% and 20% CD28 receptor blocade after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Incidence of antidrug antibodies (ADA) and neutralizing antibodies (NAb) after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Type, incidence, severity, timing, seriousness and relatedness of abnormal cytokine levels after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.

OTHER OUTCOMES:
To explore through study completion the immune activity (whole blood TruCulture® assay) of FR104 (Part 1 and 2). | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
To explore through study completion the effect of FR104 on the response to keyhole limpet hemocyanin (KLH) challenge (Part 1, Cohort B). | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
To evaluate through study completion the effect of FR104 on lymphocytes subsets (Part 1: 0.2 and 0.5 mg/kg doses [Cohort A], 2 doses up to 5 (or lower than 0.5) mg/kg [Cohort B, Groups 9 and 9 bis]) | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Apparent clearance (CL/F) after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.
Apparent volume of distribution (Vz/F) after single and two repeat iv administrations of FR104 | 4 months
  During each treatment period, subjects will be housed and monitored at the study center from the day before dosing (Day-1) until Day 5. Thenafter, each subject will attend ambulatory visit at predefined days until day 113.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ramael, Principal Investigator — SGS Antwerpen
Locations (1):
- SGS Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided